CLINICAL TRIAL: NCT04427488
Title: The Effect of Exercises Performed According to Circadian Rhythm in Type 2 Diabetes
Acronym: Circadian
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, merve yilmaz menek, Lecturer, Istanbul Medipol University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: merveymz
Record Dates: First submitted 2020-06-08; First posted 2020-06-11 (Actual); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: Type 2 Diabetes
Keywords: Circadian Rhthym; Exercise; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Morning Chronotype (MC) Group (Experimental): In the MC group, exercises were applied in the morning hours for the first 6 weeks and in the evening hours for the next 6 weeks.
  Interventions: Other: Morning Chronotype group
- Evening Chronotype (EC) Group (Experimental): The EC exercises were applied in the evening hours for the first 6 weeks and in the morning hours for the next 6 weeks
  Interventions: Other: Evening Chronotype group

INTERVENTIONS:
Other: Morning Chronotype group — Total of 12 weeks aerobic and strengthening exercises in different timing of the day.
  Arms: Morning Chronotype (MC) Group
Other: Evening Chronotype group — Total of 12 weeks aerobic and strengthening exercises in different timing of the day.
  Arms: Evening Chronotype (EC) Group

SUMMARY:
Type 2 diabetes is a metabolic disease characterized by partial insulin deficiency or insulin resistance in peripheral tissue. Type 2 diabetes, which has a very high prevalence worldwide, is a socially serious health problem. Exercise has beneficial effects on the glycemic profile, such as decreased glycemic hemoglobin (HbA1c) level, increased maximum oxygen consumption (VO2max) and improved insulin sensitivity in diabetes patients. When the literature is examined, it is seen that exercise is also effective in improving metabolic health. Although the metabolic benefits of exercise have been shown, there is no study of which type of exercise is more beneficial in what time of day in individuals with Type 2 diabetes. Circadian rhythm plays an important role in clarifying this issue because the circadian rhythm is impaired in the glucose metabolism of individuals with type 2 diabetes.The aim of this study is to investigate which exercise is more effective in which time period for individuals with Type 2 diabetes

DETAILED DESCRIPTION:
INTRODUCTION: Type 2 diabetes is a metabolic disease characterized by partial insulin deficiency or insulin resistance in peripheral tissue. Type 2 diabetes, which has a very high prevalence worldwide, is a socially serious health problem. Complications seen with the disease negatively affect human health. Physical activity and regular exercise are shown in the first place with pharmacological treatment and diet approaches in the treatment of Type 2 diabetes. Exercise has beneficial effects on the glycemic profile, such as decreased glycemic hemoglobin (HbA1c) level, increased maximum oxygen consumption (VO2max) and improved insulin sensitivity in diabetes patients. When the literature is examined, it is seen that exercise is also effective in improving metabolic health. Although the metabolic benefits of exercise have been shown, there is no study of which type of exercise is more beneficial in what time of day in individuals with Type 2 diabetes. Circadian rhythm plays an important role in clarifying this issue because the circadian rhythm is impaired in the glucose metabolism of individuals with type 2 diabetes.

AIM: The aim of this study is to evaluate the effectiveness of structured exercises given in accordance with the circadian rhythm of individuals with type 2 diabetes.

METHOD: 30 people with Type 2 diabetes in accordance with the criteria for inclusion in the Department of Endocrine and Metabolism Diseases of Medipol University Hospital in Istanbul will be included in this study. Individuals who have been diagnosed with Type 2 diabetes between the ages of 35-65, who have body mass index between 25 and 30, who have HbA1c value> 6.5%, who have fasting blood glucose>126 mg/dl, who have Type 2 diabetes between 5-10 years, who have inactive physical activity, who independently can walk and volunteer to exercise for at least 3 days a week will be included in our study. Type 1 diabetes individuals, diagnosed with Latent Autoimmune Diabetes in Adults (LADA), having diabetic Ketoacidosis coma, orthopedic or surgical problems to prevent walking and exercising, foot ulcers, individuals have any neurologıcal problem and individuals with cardiac, pulmonary or systematic diseases that will cause contraindications will not be included in the study. Blood sample evaluations, circadian rhythm evaluation, 6-minute walking test, 30-second sit to stand test, quality of life assessment with Ferrans&Powers Quality of Life Index of the individuals included will be carried out at the beginning of the study (T0) and at 6 (T1), 12 (T2) and 18 (T3) weeks after the study started Participants will be divided into two groups, morning (MC) and evening chronotypes (EC), according to their circadian rhythms. In both groups, there was a 6-week control period in which the participants continued to their routine treatment and did not perform any specific exercises. In the MC group, exercises were applied in the morning hours for the first 6 weeks and in the evening hours for the next 6 weeks. The EC exercises were applied in the evening hours for the first 6 weeks and in the morning hours for the next 6 weeks. A structured exercise program with aerobic and strengthening exercises was carried out in both groups for 3 days a week over 12 weeks. . Individuals were evaluated in terms of the blood test, functional capacity and quality of life at the baseline, 6 weeks before the exercise, 6 and 12 weeks after the exercises.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Type 2 diabetes
* Between the ages of 35-65
* Body mass index between 25 and 30
* HbA1c value> 6.5%
* Fasting blood glucose>126 mg/dl
* Inactive physical activity level
* Who independently can walk and volunteer to exercise for at least 3 days a week

Exclusion Criteria:

* Clinical diagnosis of Type 1 diabetes
* Clinical diagnosis of Latent Autoimmune Diabetes in Adults (LADA)
* Having diabetic Ketoacidosis coma
* Orthopedic or surgical problems to prevent walking and exercising
* Foot ulcers
* Neurologıcal, cardiac, pulmonary or systematic diseases

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2021-08-15 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
HbA1c evaluation | 3 hours
  Blood sample scores are changeable
Fasting glucose evaluation | 3 hours
  Blood sample are changeable
HDL (high density lipoprotein) evaluation | 3 hours
  Blood sample are changeable
LDL (low density lipoprotein) evaluation | 3 hours
  Blood sample are changeable
Total cholesterol evaluation | 3 hours
  Blood sample are changeable
Circadian Rhythm Evaluation with Morningness Eveningness Questionnaire | 10 minutes
  Scores can range from 16-86. Scores of 41 and below indicate "evening types". Scores of 59 and above indicate "morning types". Scores between 42 and 58 indicate "intermediate types" in Morningness Eveningness Questionnaire

SECONDARY OUTCOMES:
6-minute walking test | 10 minutes
  An increase in the distance walked indicates improvement in basic mobility.
30-second sit to stand test | 10 minutes
  The wide variety of ability levels indicates with high scores
Ferrans&Powers Quality of Life | 10 minutes
  High scores indicates high Quality of life in individuals with diabetes

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
An article will be published at the end of this study. IIPD can be accessed with this article.

REFERENCES:
- [Result] Savikj M, Gabriel BM, Alm PS, Smith J, Caidahl K, Bjornholm M, Fritz T, Krook A, Zierath JR, Wallberg-Henriksson H. Afternoon exercise is more efficacious than morning exercise at improving blood glucose levels in individuals with type 2 diabetes: a randomised crossover trial. Diabetologia. 2019 Feb;62(2):233-237. doi: 10.1007/s00125-018-4767-z. Epub 2018 Nov 13. PMID 30426166
- [Derived] Menek MY, Budak M. Effect of exercises according to the circadian rhythm in type 2 diabetes: Parallel-group, single-blind, crossover study. Nutr Metab Cardiovasc Dis. 2022 Jul;32(7):1742-1752. doi: 10.1016/j.numecd.2022.04.017. Epub 2022 Apr 29. PMID 35606229